CLINICAL TRIAL: NCT03605680
Title: A Phase 3, Randomized, Double-blind, Multicenter, Placebo-controlled, Parallel-group Trial Evaluating the Efficacy, Safety, and Tolerability of Centanafadine Sustained-release Tablets in Adults With Attention-deficit/Hyperactivity Disorder
Brief Title: A Trial Evaluating the Efficacy, Safety, & Tolerability of Centanafadine Sustained-release Tablets in Adults With Attention-deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 405-201-00013
Record Dates: First submitted 2018-06-28; First posted 2018-07-30 (Actual); Results first posted 2021-05-05 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Attention Deficit Disorder; Attention Deficit Hyperactivity Disorder
Keywords: Centanafadine; ADHD; ADD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 1-(naphthalen-2-yl)-3-azabicyclo(3.1.0)hexane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single-blind Run-in Period: Placebo (Experimental): Placebo-matching tablets BID (twice daily) on Day -7 through Baseline (Day -1).
  Interventions: Other: Placebo
- Double-blind Treatment Period: Centanafadine SR 200 mg (Experimental): Following Single-blind Run-in Period, participants with <30% improvement on Adult ADHD Self Report Scale (ASRS) scale score were randomized to receive centanafadine 200 mg SR tablets BID orally on Day 1 through Day 42 in the Double-blind Treatment Period.
  Interventions: Drug: Centanafadine SR
- Double-blind Treatment Period: Centanafadine SR 400 mg (Experimental): Following Single-blind Run-in Period, participants with <30% improvement on Adult ADHD Self Report Scale (ASRS) scale score were randomized to receive centanafadine 400 mg SR tablets BID orally on Day 1 through Day 42 in the Double-blind Treatment Period.
  Interventions: Drug: Centanafadine SR
- Double-blind Treatment Period: Placebo (Placebo Comparator): Following Single-blind Run-in Period, participants with <30% improvement on Adult ADHD Self Report Scale (ASRS) scale score were randomized to receive centanafadine SR matching placebo tablets BID orally on Day 1 through Day 42 in the Double-blind Treatment Period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Centanafadine SR — 100 mg, BID, oral tablets
  Other Names: EB-1020
  Arms: Double-blind Treatment Period: Centanafadine SR 200 mg
Other: Placebo — BID, oral tablet.
  Arms: Double-blind Treatment Period: Placebo; Single-blind Run-in Period: Placebo
Drug: Centanafadine SR — 200 mg, BID, oral tablets
  Other Names: EB-1020
  Arms: Double-blind Treatment Period: Centanafadine SR 400 mg

SUMMARY:
This study evaluates the efficacy, safety, and tolerability of centanafadine sustained-release tablets in adults with attention-deficit/hyperactivity disorder (ADHD). Participants will either receive a twice-daily dose of centanafadine sustained-release tablets, or twice-daily placebo.

DETAILED DESCRIPTION:
Screening & Washout Period: up to 28 days Investigational Treatment Period: 49 days Follow-up Period : 7 days or 10 days

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) criteria for ADHD (including predominantly inattentive presentation, hyperactive presentation, or combined presentation) as confirmed by the Adult ADHD Clinical Diagnostic Scale (ACDS) Version 1.2. To confirm that ADHD is the primary diagnosis, the Mini International Neuropsychiatric Interview (MINI) will be used to identify and exclude other psychiatric conditions which would preclude enrollment.
* Participants who were not receiving any pharmacological treatment for ADHD must have an Adult ADHD Investigator Symptom Rating Scale (AISRS) score of ≥ 28 at screening and baseline. Participants who were receiving pharmacological treatment for ADHD at screening must have a minimum AISRS score of ≥ 22 at screening, and a score of ≥ 28 at baseline.
* All participants must be willing to discontinue all prohibited psychotropic medications starting from the time of signing the informed consent through the 7-day follow-up period. Participants that do not rollover into Trial 405-201-00015 (NCT03605849) must be willing to discontinue all prohibited psychotropic medications starting from the time of signing the informed consent until after the follow-up telephone call 10 days after the last dose of investigational medicinal product (IMP).
* Participants must have a Clinical Global Impression-Severity of Illness Scale (CGI-S) score of ≥ 4 (≥ moderate impairment) at baseline.

Exclusion Criteria:

* Participants with a DSM-5 diagnosis of Other Specified or Unspecified Attention Deficit/Hyperactivity Disorder.
* Participants has a current comorbid psychiatric disorder that either could be expected to require treatment with medications prohibited in this trial, or to confound efficacy or safety assessments. Examples include, but are not limited to, psychotic disorder, bipolar disorder, generalized anxiety disorder, obsessive-compulsive disorder, panic disorder, a current major depressive episode, or posttraumatic stress disorder, as established by the Mini International Neuropsychiatric Interview (MINI).
* In the opinion of the investigator, participants has not derived significant therapeutic benefit from 2 or more ADHD therapies of 2 different classes (eg, amphetamine and methylphenidate) given with an acceptable dose and duration during adulthood (aged 18 or older). NOTE: If participants has not derived significant therapeutic benefit due to an inability to tolerate side effects, eligibility can be discussed on case-by-case basis with the medical monitor.
* Participants who have a positive alcohol test (via breathalyzer or blood), a positive drug screen assessed prior to the baseline visit for cocaine, other illicit drugs (including marijuana), or prescription or over-the-counter (OTC) ADHD medications will be early terminated. This includes medications such as opioids or benzodiazepines taken without prescription.
* In the opinion of the investigator, the participants is unable to adhere to the treatment regimen or other requirements outlined in the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 604 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-04-11 (Actual); Study Completion 2020-04-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 45 investigative sites in the United States from 16 January 2019 to 11 April 2020.
Pre-assignment Details: A total of 604 participants were enrolled in the study, out of which 584 were treated during the placebo Run-in Period. Out of 584, 466 participants were randomized into one of the three treatment groups (centanafadine 200 mg, centanafadine 400 mg, or placebo) in the Double-blind Treatment Period.
Groups:
- Single-blind (SB) Run-in Period: Placebo: Placebo-matching tablets BID (twice daily) on Day -7 through Baseline (Day -1).
- Double-blind Treatment Period: Centanafadine SR 200 mg: Following Single-blind Run-in Period, participants with <30% improvement on Adult ASRS scale score were randomized to receive centanafadine 200 mg SR tablets BID orally on Day 1 through Day 42 in the Double-blind Treatment Period.
- Double-blind Treatment Period: Centanafadine SR 400 mg: Following Single-blind Run-in Period, participants with <30% improvement on Adult ASRS scale score were randomized to receive centanafadine SR 200 mg tablets BID orally on Day 1 through Day 7 and were then escalated to their target total daily dose (TDD) of centanafadine 400 mg on Day 8 through Day 42 in the Double-blind Treatment Period.
- Double-blind Treatment Period: Placebo: Following Single-blind Run-in Period, participants with <30% improvement on ASRS scale score were randomized to receive centanafadine matching placebo SR tablets BID orally on Day 1 through Day 42 in the Double-blind Treatment Period.
Period: SB Placebo Run-in Period (1 Week)
Arm/Group | Single-blind (SB) Run-in Period: Placebo | Double-blind Treatment Period: Centanafadine SR 200 mg | Double-blind Treatment Period: Centanafadine SR 400 mg | Double-blind Treatment Period: Placebo
Started | 604 | 0 | 0 | 0
Treated | 584 | 0 | 0 | 0
Completed | 466 | 0 | 0 | 0
Not Completed | 138 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 0 | 0 | 0
Not completed — Non-compliance With Study Drug | 3 | 0 | 0 | 0
Not completed — Protocol Deviation | 13 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 0 | 0 | 0
Not completed — Site Terminated by Sponsor | 1 | 0 | 0 | 0
Not completed — Physician Decision | 6 | 0 | 0 | 0
Not completed — Reason not Specified | 87 | 0 | 0 | 0
Period: Double-blind Treatment Period (6 Weeks)
Arm/Group | Single-blind (SB) Run-in Period: Placebo | Double-blind Treatment Period: Centanafadine SR 200 mg | Double-blind Treatment Period: Centanafadine SR 400 mg | Double-blind Treatment Period: Placebo
Started | 0 | 154 | 156 | 156
Completed | 0 | 110 | 117 | 121
Not Completed | 0 | 44 | 39 | 35
Not completed — Randomized but Not Treated in Double-Blind Treatment Period | 0 | 5 | 7 | 8
Not completed — Adverse Event | 0 | 8 | 8 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 3 | 4 | 3
Not completed — Non-compliance with Study Drug | 0 | 3 | 1 | 2
Not completed — Protocol Deviation | 0 | 14 | 7 | 5
Not completed — Withdrawal by Subject | 0 | 4 | 4 | 7
Not completed — Physician Decision | 0 | 1 | 2 | 0
Not completed — Reason not Specified | 0 | 5 | 4 | 3
Not completed — Reason due to COVID-19 | 0 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Participants who participated only in the Run-in Period and Full Analysis Set (FAS) including all participants in the safety sample who had a Baseline value and at least one valid post-randomization efficacy evaluation for adult ADHD investigator symptom rating scale (AISRS) total score in the Double-blind Treatment Period.
Groups:
- Placebo: Single-blind Run-in Period Only: Placebo-matching tablets BID (twice daily) on Day -7 through Baseline (Day -1) in the Run-in Period only. Participants did not continue to Double-blind Treatment Period.
- Double-blind Treatment Period: Placebo + Centanafadine SR 200 mg: Participants received centanafadine SR matching placebo tablets in Single-blind Run-in Period. Participants who showed >=30% improvement in Adult ASRS at Baseline were early terminated and the remaining participants were randomized to receive centanafadine SR 200 mg tablets BID orally on Day 1 through Day 42 in the Double-blind Treatment Period.
- Double-blind Treatment Period: Placebo + Centanafadine SR 400 mg: Participants received centanafadine SR matching placebo tablets in Single-blind Run-in Period. Participants who showed >=30% improvement in Adult ASRS at Baseline were early terminated and the remaining participants were randomized to receive centanafadine SR 200 mg tablets BID orally on Day 1 through Day 7 and were then escalated to their target TDD of centanafadine 400 mg on Day 8 through Day 42 in the Double-blind Treatment Period.
- Double-blind Treatment Period: Placebo + Placebo: Participants received centanafadine SR matching placebo tablets in Single-blind Run-in Period. Participants who showed >=30% improvement in Adult ASRS at Baseline were early terminated and the remaining participants were randomized to receive centanafadine SR matching placebo tablets BID orally on Day 1 through Day 42 in the Double-blind Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Placebo: Single-blind Run-in Period Only | Double-blind Treatment Period: Placebo + Centanafadine SR 200 mg | Double-blind Treatment Period: Placebo + Centanafadine SR 400 mg | Double-blind Treatment Period: Placebo + Placebo | Total
Number analyzed (Participants) | 138 | 154 | 156 | 156 | 604
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (9.4) | 36.6 (9.8) | 35.3 (10.4) | 35.0 (9.9) | 35.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 76 | 75 | 76 | 284
  Male | 81 | 78 | 81 | 80 | 320
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 34 | 38 | 29 | 129
  Not Hispanic or Latino | 110 | 119 | 116 | 124 | 469
  Unknown or Not Reported | 0 | 1 | 2 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 3 | 0 | 4
  Asian | 5 | 4 | 2 | 4 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 0 | 3
  Black or African American | 22 | 19 | 23 | 21 | 85
  White | 107 | 126 | 123 | 130 | 486
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 4 | 1 | 11
Adult Attention-deficit/Hyperactivity Disorder (ADHD) Investigator Symptom Rating Scale (AISRS) [Mean (Standard Deviation); unit: score on a scale] — The Adult Investigator Symptom Rating Scale (AISRS) is an 18-item clinician rating scale to evaluate individual ADHD symptoms on a scale of 0 (none) to 3 (severe). The total sum ranges from 0 (no ADHD symptoms) to 54 (extremely severe ADHD symptoms). Population: Data for ADHD AISRS scale was collected only for Double-blind Treatment Period arms.
  score on a scale
    number analyzed (Participants) | 0 | 154 | 156 | 156 | 466
    (all) |  | 39.7 (6.7) | 39.4 (6.8) | 39.4 (7.1) | 39.5 (6.8)
Clinical Global Impression-Severity of Illness Scale (CGI-S) [Mean (Standard Deviation); unit: score on a scale] — CGI-S is an observer-rated scale used to measure symptom severity with a total score range of 0 to 7 where 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants. Population: Data for CGI-S scale was collected only for Double-blind Treatment Period arms. Number analyzed is the number of participants with data available for analyses.
  score on a scale
    number analyzed (Participants) | 0 | 153 | 156 | 156 | 465
    (all) |  | 4.5 (0.6) | 4.5 (0.6) | 4.5 (0.6) | 4.5 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in ADHD Investigator Symptom Rating Scale (AISRS)
Description: The Adult Investigator Symptom Rating Scale (AISRS) is an 18-item clinician rating scale to evaluate individual ADHD symptoms on a scale of 0 (none) to 3 (severe). The total sum ranges from 0 (no ADHD symptoms) to 54 (extremely severe ADHD symptoms). Negative change from Baseline indicates improvement. Mixed-effect model repeated measure (MMRM) was used for analysis.
Time Frame: Baseline and Day 42
Population: Efficacy sample FAS included all participants in the safety sample who had a Baseline value and at least one valid post-randomization efficacy evaluation for AISRS total score in the Double-blind Treatment Period. Overall number analysed are the participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Double-blind Treatment Period: Centanafadine SR 400 mg: Following Single-blind Run-in Period, participants with <30% improvement on Adult ASRS scale score were randomized to receive centanafadine SR 200 mg tablets BID orally on Day 1 through Day 7 and were then escalated to their target TDD of centanafadine 400 mg on Day 8 through Day 42 in the Double-blind Treatment Period.
- Double-blind Treatment Period: Placebo: Following Single-blind Run-in Period, participants with <30% improvement on Adult ASRS scale score were randomized to receive centanafadine matching placebo SR tablets BID orally on Day 1 through Day 42 in the Double-blind Treatment Period.
Arm/Group | Double-blind Treatment Period: Centanafadine SR 200 mg | Double-blind Treatment Period: Centanafadine SR 400 mg | Double-blind Treatment Period: Placebo
Number analyzed (Participants) | 147 | 147 | 144
score on a scale | -10.1 (0.99) | -9.73 (0.98) | -6.98 (0.98)
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Centanafadine SR 200 mg vs Double-blind Treatment Period: Placebo; Test type: Superiority; p = 0.0193, MMRM; Least Squares (LS ) Mean Difference = -3.15, 95% CI 2-sided [-5.79 to -0.51]; The comparison between the centanafadine and the placebo group was tested at a significance level of 0.05
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Centanafadine SR 400 mg vs Double-blind Treatment Period: Placebo; Test type: Superiority; p = 0.0392, MMRM; LS Mean Difference = -2.74, 95% CI 2-sided [-5.35 to -0.14]

2. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity of Illness Scale (CGI-S)
Description: CGI-S is an observer-rated scale used to measure symptom severity with a total score range of 0 to 7 where 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants. A negative change from Baseline indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline and Day 42
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Double-blind Treatment Period: Centanafadine SR 200 mg | Double-blind Treatment Period: Centanafadine SR 400 mg | Double-blind Treatment Period: Placebo
Number analyzed (Participants) | 146 | 147 | 144
score on a scale | -0.78 (0.09) | -0.79 (0.08) | -0.52 (0.08)
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Centanafadine SR 200 mg vs Double-blind Treatment Period: Placebo; Test type: Superiority; p = 0.0232, MMRM; LS Mean Difference = -0.27, 95% CI 2-sided [-0.50 to -0.04]; The comparison between the centanafadine and the placebo group was tested at a significance level of 0.05
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Centanafadine SR 400 mg vs Double-blind Treatment Period: Placebo; Test type: Superiority; p = 0.0162, MMRM; LS Mean Difference = -0.28, 95% CI 2-sided [-0.51 to -0.05]; The comparison between the centanafadine and the placebo group was tested at a significance level of 0.05

3. Other Pre Specified Outcome: Adverse Event Reporting
Description: Frequency and severity of treatment-emergent adverse events (TEAEs) will be assessed to determine safety and tolerability of centanafadine SR tablets.
Time Frame: Up to 59 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: ADHD Impact Module - Adult (AIM-A)
Description: Scale composed of 3 subscales with a maximum score of 100. A lower score indicates a worse outcome. Exploratory endpoint; comparison of baseline score to other points throughout the study.
Time Frame: Up to 42 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Adult ADHD Self Report Scale (ASRS)
Description: An 18 question report, total score ranges from 0 to 124. A higher score denotes a worse outcome. Exploratory endpoint; comparison of baseline score to other points throughout the study.
Time Frame: Up to 42 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Adult ADHD Investigator Symptom Rating Scale (AISRS)
Description: Change from baseline total score compared to every scheduled visit. Each subscale is composed of 9 items each. Scores can range from 0 to 27, with a higher score representing a worse outcome. Change from baseline scores are compared to every scheduled visit score.
Time Frame: Up to 42 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 59 days
Description: Safety sample included randomized participants who received at least 1 dose of study drug. The Placebo: Single-blind Run-in Period Only arm includes AEs that occurred during single-blind run-in period for participants who received at least 1 dose of study drug but did not participate in DB period. As pre-specified in SAP, AEs that occurred in Single-blind Placebo Run-In period for participants who received treatment in DB period was reported in DB treatment arms based on DB treatment received.
Groups:
- Placebo: SB Run-in Period Only: Placebo-matching tablets BID (twice daily) on Day -7 through Baseline (Day -1) in the Single-blind Run-in Period only. Participants did not continue to Double-blind Treatment Period.
- Placebo + Centanafadine SR 200 mg: Participants received centanafadine SR matching placebo tablets in Single-blind Run-in Period. Participants who showed >=30% improvement in ASRS at Baseline were early terminated and the remaining participants were randomized to receive centanafadine SR 200 mg tablets BID orally on Day 1 through Day 42 in the Double-blind Treatment Period.
- Placebo + Centanafadine SR 400 mg: Participants received centanafadine SR matching placebo tablets in Single-blind Run-in Period. Participants who showed >=30% improvement in ASRS at Baseline were early terminated and the remaining participants were randomized to receive centanafadine SR 200 mg tablets BID orally on Day 1 through Day 7 and were then escalated to their target TDD of centanafadine 400 mg on Day 8 through Day 42 in the Double-blind Treatment Period.
- Placebo + Placebo: Participants received centanafadine SR matching placebo tablets in Single-blind Run-in Period. Participants who showed >=30% improvement in ASRS at Baseline were early terminated and the remaining participants were randomized to receive centanafadine SR matching placebo tablets BID orally on Day 1 through Day 42 in the Double-blind Treatment Period.
Arm/Group | Placebo: SB Run-in Period Only | Placebo + Centanafadine SR 200 mg | Placebo + Centanafadine SR 400 mg | Placebo + Placebo
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/149 | 0/149 | 0/148
Serious Adverse Events (participants affected / at risk) | 0/138 | 2/149 | 0/149 | 0/148
Other Adverse Events (participants affected / at risk) | 2/138 | 25/149 | 22/149 | 18/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: SB Run-in Period Only (N=138) | Placebo + Centanafadine SR 200 mg (N=149) | Placebo + Centanafadine SR 400 mg (N=149) | Placebo + Placebo (N=148)
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: SB Run-in Period Only (N=138) | Placebo + Centanafadine SR 200 mg (N=149) | Placebo + Centanafadine SR 400 mg (N=149) | Placebo + Placebo (N=148)
Dry Mouth (Gastrointestinal disorders) | 0 | 6 | 9 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 8 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 9 | 11 | 2
Headache (Nervous system disorders) | 2 | 5 | 7 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT03605680/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/80/NCT03605680/SAP_001.pdf